CLINICAL TRIAL: NCT05143528
Title: A Multicenter, Phase III, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Nilotinib BE in Subjects With Early Alzheimer's Disease (NILEAD)
Brief Title: Evaluating the Efficacy and Safety of Nilotinib BE in Subjects With Early Alzheimer's Disease
Acronym: NILEAD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KeifeRx, LLC (Industry)
Collaborators: Worldwide Clinical Trials (Other); Life Molecular Imaging GmbH (Industry); Sun Pharmaceuticals Industries Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFRX 2021
Record Dates: First submitted 2021-11-02; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer Disease
Keywords: early Alzheimer's disease; CDR; Amyloid PET; CSF Amyloid; Volumetric MRI; TAU PET
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Double-Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Placebo (Placebo Comparator): 425 subjects will be randomized to the placebo group.
  Interventions: Drug: Placebo
- Arm B: Experimental Low Dose (Active Comparator): 425 subjects to each of the Nilotinib BE, 84mg.
  Interventions: Drug: Nilotinib BE 84mg
- Arm C: Experimental High Dose (Active Comparator): 425 subjects to each of the Nilotinib BE, 112mg.
  Interventions: Drug: Nilotinib BE 112 mg

INTERVENTIONS:
Drug: Nilotinib BE 84mg — 84 mg capsule
  Arms: Arm B: Experimental Low Dose
Drug: Nilotinib BE 112 mg — 112 mg capsule
  Arms: Arm C: Experimental High Dose
Drug: Placebo — placebo capsule
  Arms: Arm A: Placebo

SUMMARY:
This study will investigate the safety and efficacy of a Tyrosine Kinase Inhibitor (TKI) called Nilotinib BE (bioequivalent) in individuals with Early Alzheimer's disease (EAD). This is a multi-center double blinded, Phase 3 study, that will enroll patients for three years in approximately 50 centers nationwide. The total duration of the study will be for five years.

DETAILED DESCRIPTION:
Number of Subjects: Approximately 1275 subjects will be randomized 1:1:1 across Nilotinib BE, 84mg or 112mg or matching placebo

Number of Centers: Approximately 50 centers US-Wide

Duration of Study: Enrollment will be (competitive) opened for 3 years (36 months) and total study duration is approximately 5 years

Core Study: Approximately 425 subjects will be randomized to the placebo group (arm A) and 425 subjects to each of the Nilotinib BE, 84mg (arm B) and 112mg (arm C) groups.

Biomarker Sub-study: Approximately 180 subjects (60 subjects per group) will be randomized for the CSF biomarker sub-study at Baseline and 18 months (Week 72).

Approximately 164 subjects (48 per group) will be randomized to the imaging sub-studies, including amyloid PET, tau PET and vMRI, at Baseline and 18 months (week 72).

Eligible subjects are diagnosed with dementia due to AD according to the National Institute of Aging-Alzheimer's Association (NIA-AA) core clinical criteria for early AD. Participants must have a global CDR score of 0.5 to 1.0 and a CDR Memory Box score of 0.5 or greater at Screening and Baseline and/or MMSE score greater than or equal to 20 at Screening and Baseline and less than or equal to 27 at Screening and Baseline. Male or female subjects aged ≥55 and ≤ 85 years, at the time of IC.

ELIGIBILITY:
Inclusion Criteria:

* 1- Diagnosis of dementia due to AD

  2- Meet the National Institute of Aging-Alzheimer's Association (NIA-AA) core clinical criteria for dementia due to AD

  3- Have a global CDR score of 0.5 to 1.0 and a CDR Memory Box score of 0.5 or greater at Screening and Baseline

  4- Have an MMSE score greater than or equals to 20 at Screening and less than or equals to 27 at Screening and Baseline

  5- Have a positive amyloid PET (visual reading) or positivity threshold of CSF Aβ[1-42] < 660ng/ml or ptau/Aβ[1-42] >0.09 using INNOTEST Enzyme-Linked ImmunoAssay (ELISA) technique (Fujirebio, Ghent, Belgium).

  6- QTc (corrected Q wave to the end of the T wave) interval 350-480 ms, inclusive for both men and women

  7- English or Spanish fluency

  8- Report a history of subjective memory decline with gradual onset and slow progression over the last 1 year before Screening; must be corroborated by an informant

  9- Positive biomarker for brain amyloid pathology as indicated by at least 1 of the following:
  1. PET assessment of imaging agent uptake into brain
  2. CSF assessment of Aβ[1-42] or ptau/Aβ[1-42] NOTE: To confirm eligibility, a positive amyloid result is needed in only 1 of the 2 procedures, including PET or CSF measurement.

     10- Male or female subjects aged ≥55 and ≤ 85 years, at the time of informed consent (IC)

     11- Body mass index (BMI) greater than 17 and less than 35 at Screening

     12- If receiving an approved AD treatment, such as acetylcholinesterase inhibitors (AChEIs), or memantine, or both for AD, must be on a stable dose for at least 12 weeks prior to Baseline. Treatment-naïve subjects for AD can be entered into the study. Unless otherwise stated, subjects must have been on stable doses of all other (i.e., non-AD-related) permitted concomitant medications for at least 4 weeks prior to Baseline.

     13- Have an identified study partner. The study partner must provide separate written IC. In addition, this person must be willing and able to provide follow-up information on the subject throughout the course of the study. This person must, in the opinion of the investigator, spend sufficient time with the subject on a regular basis such that the study partner can reliably fulfill the study requirements. A permanent study partner need not be living in the same residence with the subject. For such a study partner not residing with the subject, the investigator has to be satisfied that the subject can contact the study partner readily during the times when the study partner is not with the subject. Study partners need to participate in person for visits where clinical assessment of CDR (global and CDR-SB), ADAS-Cog, ADCS-ADL-MCI and NPI.

     14- Provide written IC. If a subject lacks capacity to consent in the investigator's opinion, the subject's assent should be obtained, if required in accordance with local laws, regulations and customs, plus the written IC of a legal representative should be obtained.

     15- Willing and able to comply with all aspects of the protocol.

Biomarker Sub-study

NOTE: Subjects may consent to either one or both the PET and CSF assessments, but to confirm eligibility, a positive amyloid result is needed in only 1 of the 2 procedures (Amyloid PET (via visual reading) or CSF assessment). The historical imaging data and CSF assessment results must be made available to the sponsor or medical monitor to confirm amyloid positivity and eligibility.

Historical PET and CSF assessments will ONLY be used for determination of eligibility. However, subjects who enroll in the biomarker sub study MUST participate in one or more of the amyloid and tau PET, vMRI and CSF assessments according to the Assessments Schedule in the sponsor protocol.

Patients may use any amyloid PET tracer to prove eligibility, but they must use only the sponsor provided tracer at Baseline and End of Treatment- unless the same tracer was used within 12 months from Baseline and the data can be provided to the investigator and the subject has not participated in any subsequent anti-amyloid study or treatment.

Exclusion Criteria:

1. Subjects who are on anti-amyloid therapy (i.e. vaccine or antibody) or who were receiving anti-amyloid vaccines (i.e. aducunamab) or anti-tau vaccines less than 3 months before Screening.
2. Women of childbearing potential (WCBP). NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
3. Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the subject's AD.
4. Any psychiatric diagnosis or symptoms, (e.g., hallucinations, major depression, or delusions) that could interfere with study procedures in the subject.
5. Geriatric Depression Scale (GDS) score greater than or equal to 8 at Screening.
6. Contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (e.g., in skull and cardiac devices other than those approved as safe for use in MRI scanners).
7. Evidence of other clinically significant lesions on brain MRI that could indicate a dementia diagnosis other than AD.
8. Other significant pathological findings on brain MRI, including but not limited to: more than 4 micro hemorrhages (defined as 10mm or less at the greatest diameter); a single macro hemorrhage greater than 10mm at greatest diameter; an area of superficial siderosis; evidence of vasogenic edema; evidence of cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions; evidence of multiple lacunar infarcts or stroke involving a major vascular territory, severe small vessel, or white matter disease; space occupying lesions; or brain tumors (however, lesions diagnosed as meningiomas or arachnoid cysts and less than 1cm at their greatest diameter need not be exclusionary).
9. Patients with hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥481 ms
10. Concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infraction or cardiac failure, angina, arrhythmia
11. Presence of cardiac conditions including:

    1. Cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke)
    2. Congestive heart failure
    3. Second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
    4. Any history of Torsade de Pointes
12. Treatment with any of the following drugs at the time of Screening or the preceding 30 days, and/or planned use over the course of the trial:

    1. Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine)
    2. Treatment with QT prolonging drugs (www.crediblemeds.org)- excluding Selective Serotonin Reuptake Inhibitors (SSRIs) (e.g. Citalopram, Paxil, Zoloft, Cymbalta, Sertraline, etc...)
    3. Strong CYP3A4 inhibitors (including grapefruit juice). The concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) must be avoided. Grapefruit products may also increase serum concentrations of Nilotinib (Tasigna). Should treatment with any of these agents be required, therapy with Nilotinib BE should be interrupted.
    4. Anticoagulants, including Coumadin (warfarin), heparin, enoxaparin, daltiparin, xarelto, etc.
13. St. John's Wort and the concomitant use of strong other CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) must be avoided since these agents may reduce the concentration of Nilotinib.
14. Any immunological disease which is not adequately controlled, or which requires treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives of monoclonal antibodies), systemic immunosuppressant's, or plasmapheresis during the study.
15. Subjects with a bleeding disorder that is not under adequate control (including a platelet count <50,000 or international normalized ratio [INR] >1.5 for subjects who are not on anticoagulant treatment, e.g., warfarin). Subjects who are on anticoagulant therapy should have their anticoagulant status optimized and be on a stable dose for 4 weeks before Screening.
16. Have thyroid stimulating hormone above normal range. Other tests of thyroid function with results outside the normal range should only be exclusionary if they are considered clinically significant by the investigator. This applies to all subjects whether or not they are taking thyroid supplements.
17. Abnormally low serum vitamin B12 levels for the testing laboratory (if subject is taking vitamin B12 injections, level should be at or above the lower limit of normal [LLN] for the testing laboratory).
18. Known to be human immunodeficiency virus (HIV) positive.
19. Any other clinically significant abnormalities in physical examination, vital signs, laboratory tests, or ECG at Screening or Baseline which in the opinion of the investigator require further investigation or treatment or which may interfere with study procedures or safety.
20. Subjects with malignant neoplasms within 3 years of Screening (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male subjects). Subjects who had malignant neoplasms but who have had at least 3 years of documented uninterrupted remission before Screening need not be excluded.
21. Answer "yes" to C-SSRS suicidal ideation Type 4 or 5, or any suicidal behavior assessment within 6 months before Screening, at Screening, or at the Baseline Visit, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening.
22. Known or suspected history of drug or alcohol abuse or dependence within 2 years before Screening.
23. Any other medical conditions (e.g., cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments.
24. Subjects who are taking prohibited medications.
25. Participation in a clinical study involving any anti-amyloid therapies (including any monoclonal antibody therapies and any β-site amyloid precursor protein cleaving enzyme [BACE] inhibitor therapies) unless it can be documented that the subject only received placebo.
26. Subjects who were dosed in a clinical study involving any new chemical entities for AD within 3 months prior to Screening unless it can be documented that the subject only received placebo.
27. Participated in any other investigational medication or device study in the 8 weeks or 5 half-lives (whichever is longer) of the medication before randomization unless it can be documented that the subject only received placebo.
28. Planned surgery which requires general anesthesia that would take place during the study. Planned surgery which requires only local anesthesia and which can be undertaken as day case without inpatient stay postoperatively need not result in exclusion if in the opinion of the investigator this operation does not interfere with study procedures and subject safety.
29. Severe visual or hearing impairment that would prevent the subject from performing psychometric tests accurately.
30. Any concomitant medication or medication excluded that could put subject at risk, or interfere with study evaluations
31. Exclusion criteria specific for the biomarker sub-study:

    * Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1275 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score at Week 72 [ Time Frame: Baseline, Week 72] | 72 weeks
  CDR-SB integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following a systematic patient examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. Prespecified severity anchors range from none = 0, questionable = 0.5, mild = 1, moderate = 2 to severe = 3 (the personal care domain omits the 0.5 score). "Sum of boxes" scoring methodology sums the score for each of the 6 domains and provides a value ranging from 0 to 18 that can change in increments of 0.5 or greater. Higher scores indicate greater disease severity. A positive change from baseline indicates clinical decline.

SECONDARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (14 Items) (ADAS-Cog 14) at Week 72 | 72 weeks
  ADAS-Cog14 comprises both cognitive tasks and clinical ratings of cognitive performance. The scale items capture word recall, ability to follow commands, the ability to correctly copy or draw an image, naming, the ability to interact with everyday objects, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. The total score ranges from 0 to 90.
  An increase in score over time indicates increasing cognitive impairment. A positive change from baseline indicates clinical decline.
Change From Baseline in Mini Mental State Examination (MMSE) Score at Week 72 | 72 weeks
  The MMSE is a widely used performance-based test of global cognitive status. It consists of 11 tasks that assess orientation, word recall, attention and calculation, language abilities, and visuospatial functions. The scores from the 11 tests are combined to obtain the total score, which ranges from 0 to 30, with lower scores over time indicating increasing cognitive impairment.
  A negative change from baseline indicates clinical decline.
Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment Version) (ADCS-ADL-MCI) Score at Week 72 | 72 weeks
  The ADCS-ADL-MCI consists of 17 instrumental items (e.g., shopping, preparing meals, using household appliances) and 1 basic item (getting dressed). Ratings reflect caregiver observations about the patient's actual functioning over the previous month and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 53, with lower values over time reflecting functional deterioration.
  A negative change from baseline indicates clinical decline.
Blood and Cerebrospinal Fluid Biomarkers | 72 weeks.
  To determine the effects of Nilotinib BE compared to placebo on blood and cerebrospinal fluid (CSF) biomarkers of AD pathology (including but not limited to amyloid beta monomer from amino acid 1 to 42 (Aβ[1-42]), Aβ monomer from amino acid 1 to 40 (Aβ[1-40]), total tau [t-tau], and phosphorylated-tau [p-tau]) at Baseline and 72 weeks.
Tau PET imaging | 72 weeks.
  To determine whether Nilotinib BE is superior to placebo in reducing brain Tau levels as measured by Tau PET using standardized uptake value ratios (SUVRs) at Baseline and 18 months (Week 72) of treatment.
Amyloid brain burden | 72 weeks
  To determine whether Nilotinib BE is superior to placebo in reducing brain amyloid levels as measured by amyloid PET using standardized uptake value ratios (SUVRs) at Baseline and 18 months (Week 72) of treatment.
Alzheimer's Disease COMposite Score (ADCOMS) | 72 weeks
  ADCOMS is a composite score comprised of ADAS-cog (4 items), MMSE (2 items) and CDR-SB (6 items). Clinical data were utilized from multiple MCI studies to develop a new score that would demonstrate maximum responsiveness to progression and to treatment in an MCI population and that would also perform well in a mild AD dementia population. A partial least squares (LS) regression model used placebo data from 4 MCI studies over 12 months to select the combination of cognitive and functional items which is most sensitive to change over time, using items from a variety of well-established and validated scales. This score assesses both cognitive and functional domains and can be offered as a single primary clinical endpoint.

OTHER OUTCOMES:
Correlation of cognitive outcomes and Amyloid PET | 72 weeks
  To evaluate the relationship between changes in amyloid PET imaging and clinical changes as measured by CDR-SB in subjects with EA.
Correlation between Amyloid and Tau with cognitive and functional outcomes | 72 weeks
  To evaluate the relationship between changes in amyloid PET imaging and other clinical changes (ADAS-cog 14, ADCS-ADL-MCI, ADCOMS and MMSE) in subjects with EAD.
  To determine whether Nilotinib BE is superior to placebo on brain tau pathology at Baseline and 18 months as measured by tau PET in subjects with EAD.

IPD SHARING:
Plan to Share IPD: Yes
KeifeRx will make all data available to the scientific community and participants and all regulatory bodies including FDA and IRB in a timely manner.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months after unblinding of the data and for a duration of 10 years.
Access Criteria: Correspondence with the Sponsor.

REFERENCES:
- [Background] Turner RS, Hebron ML, Lawler A, Mundel EE, Yusuf N, Starr JN, Anjum M, Pagan F, Torres-Yaghi Y, Shi W, Mulki S, Ferrante D, Matar S, Liu X, Esposito G, Berkowitz F, Jiang X, Ahn J, Moussa C. Nilotinib Effects on Safety, Tolerability, and Biomarkers in Alzheimer's Disease. Ann Neurol. 2020 Jul;88(1):183-194. doi: 10.1002/ana.25775. Epub 2020 May 28. PMID 32468646
- See also: Nilotinib Effects on Safety, Tolerability, and Biomarkers in Alzheimer's Disease — https://pubmed.ncbi.nlm.nih.gov/32468646/